CLINICAL TRIAL: NCT05696301
Title: Interest of Tecartherapy on a Painful Caesarean Section Scar: a Randomized Clinical Trial.
Acronym: NOCEPAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Our low recruitment is related to the fact that few women are in pain in our department 6 to 8 weeks postpartum. It was therefore decided not to extend this study.
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOI 2021 VENDITTELLI; 2022-A01492-41 (Other: 2022-A01492-41)
Record Dates: First submitted 2023-01-12; First posted 2023-01-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Cesarean Section; Postpartum; Abdominal Pain; Morbidity
Keywords: Maternal morbidity; Pain after a cesarean delivery; Postpartum care; Postnatal care
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventionnal Group (Experimental): These women will receive Tecar by Winback® technology [CE medical 1984, Norma 60601-2, ISO9001, ISO13485, CET 400 VA and RET 100 Watts, weight 4 Kg]. Each session will last for 20 minutes, and each individual will have 3 sessions over a period of 3 weeks
  Interventions: Device: Winback® on; Behavioral: self-massage of the scar
- Control (Sham Comparator): The women will follow the same study design as the experimental group with activation of the portable placebo device identical to the active medical . Each session will last for 20 minutes, and each individual will have 3 sessions over a period of 3 weeks.
  Interventions: Device: Winback® off; Behavioral: self-massage of the scar

INTERVENTIONS:
Device: Winback® on — For this study, we will use only the instrumental mode and the 4-cm electrodes. During each session, this electrode will be moved over the entire scar, with the contact between electrode and the skin provided by an adequate quantity of conductive cream.
  We will use the following 3 modes: CET, CET Dynamic, and RET; these allow us to standardize the treatment without taking into account either the thickness of the abdominal wall or the woman's morphology.
  Each session will take 20 minutes (CET for 4 min, CET Dynamic 6 min, RET 6 min and CET 4 min). The intensity of CET and RET will be adapted to each woman and the diathermy chosen according to the woman's threshold of comfort, to be determined by her at each session.
  There will be 1 session a week for 3 weeks. Portable instrument is activated.
  Arms: Interventionnal Group
Device: Winback® off — For this study, we will use only the instrumental mode and the 4-cm electrodes. During each session, this electrode will be moved over the entire scar, with the contact between electrode and the skin provided by an adequate quantity of conductive cream.
  We will use the following 3 modes: CET, CET Dynamic, and RET; these allow us to standardize the treatment without taking into account either the thickness of the abdominal wall or the woman's morphology.
  Each session will take 20 minutes (CET for 4 min, CET Dynamic 6 min, RET 6 min and CET 4 min). The intensity of CET and RET will be adapted to each woman and the diathermy chosen according to the woman's threshold of comfort, to be determined by her at each session.
  There will be 1 session a week for 3 weeks. Portable instrument is not activated.
  Arms: Control
Behavioral: self-massage of the scar — The women in both groups will have the standard recommended treatment: manual self-massage of the scar. Women's instruction in this self-massage will be structured and identical for both groups, including the provision of an informational document describing how to perform the massage. This training will be provided immediately after randomization and before the intervention or control measures.

SUMMARY:
Cesareans are a frequent procedure in obstetrics and 15.4% (95% CI, 9.9-20.9%) of women with cesareans still have pain at 3 months after delivery. Currently, self-massage of the scar is recommended to them. Post-cesarean pain is associated with psychological disorders (including, e.g., anxiety, depression). Tecar therapy could improve the healing and pain associated with cesareans and therefore improve women's quality of life and their satisfaction.

Objectives: The principal objective is to study the analgesic efficacy of tecar therapy for postoperative scar pain and/or discomfort at 3 month after cesarean delivery, by comparing it with sham tecar therapy.

A randomized clinical trial with 2 parallel arms and single blinding, to study the efficacy of this medical device for therapeutic purposes. In both groups (randomization stratified as a first cesarean or repeat cesarean), the women will have the standard recommended treatment - manual self-massage of the scar. Women's instruction in this self-massage will be structured and identical for both groups, including the provision of an informational document describing how to perform this massage. The training will be provided immediately after randomization.

* Description of the experimental group These women will receive Tecar through Winback® technology [CE medical 1984, Norma 60601-2, ISO9001, ISO13485. Class IIa medical device, CET (capacitative mode) 400 VA and RET (resistant mode) 100 Watts, weight 4 Kg)]. Each session will last for 20 minutes, and each individual will have 3 sessions over a period of 3 weeks.
* Description of the control group ("sham treatment") The women will follow the same study design as the experimental group with activation of the portable placebo device identical to the active medical. Each session will last for 20 minutes, and each individual will have 3 sessions over a 3-week period.

Principal endpoint: Visual analogic scale (VAS) for pain and/or discomfort at 3 months after delivery partum (with a ruler scored from 0 for no pain to 10 for the worst pain imaginable).

Succinct description of the products: "Tecar" is an acronym for a type of therapy (transfer electrical capacitive and resistive). The Winback® is a portable, easy-to-handle noninvasive regenerator. This study will use only the instrumental mode and 4-cm electrodes. During each session, this electrode will be moved over the entire scar. We will use the following 3 modes: capacitive (CET), CET Dynamic, and resistant (RET). These allow us to standardize the treatment without taking into account either the thickness of the abdominal wall or the woman's morphology. Each session will take 20 minutes (CET for 4 min, CET Dynamic 6 min, RET 6 min and CET 4 min). The intensity of CET and RET will be adapted to each woman and the diathermy chosen according to the woman's threshold of comfort, to be determined by her at each session, in the experimental group. There will be 1 session a week for 3 weeks.

Study plan and procedures: The eligible women will be identified by the physicians in both of the obstetrics departments participating in this study. The women will receive oral information as well as written information. If they are interested, they will be offered an inclusion visit, normally scheduled for one week later. After a second verification of the eligibility criteria at this inclusion meeting, reading the information form and signing the consent, they will be randomized into one of the two groups by random drawing. Each woman will have 3 sessions (1 session a week for 20 min for 3 consecutive weeks): active treatment by tecar therapy or sham/placebo tecar therapy. They will receive self-administered questionnaires at 3 and 6 months after delivery to be completed and returned.

DETAILED DESCRIPTION:
* Study design: A randomized clinical trial with 2 parallel arms and single blinding to study the efficacy of this medical device for therapeutic purposes.
* Procedure for early withdrawal from the treatment:

A woman can withdraw from the study early for the following reasons:

* intercurrent disease interfering with the study organization and normal protocol procedures (i.e., prolonged hospitalization for a disorder other than gynecologic or obstetric),
* death,
* the woman's decision,
* a major protocol deviation,
* and loss to follow-up (a subject lost to follow-up is a participant who did not come to the visit planned in the protocol and for whom we lack information on which we could base a judgment. It is essential to attempt by all reasonable means to obtain information and learn the reason why these women withdrew from the trial. "Lost to follow-up" will be invoked only when the investigation has been unsuccessful).

The trial may be stopped temporarily or permanently for the following reasons:

* Recruitment too low or nonexistent,
* Impossibility of obtaining funding for the trial,
* Any directive by competent authorities requiring the temporary or permanent end of the trial,
* Decision of the sponsor and of the investigator-coordinator.

  * Methods of recruitment Physician, in both obstetrics departments in which the study is planned will inform the women of the study during their postnatal consultation, planned by statute in France at 6 to 8 weeks after delivery. They will also be informed by posters displayed in the consultation sector of the two obstetrics departments.

If they are willing, they will be offered the opportunity to participate in the study; if so, a telephone appointment will be arranged for re-verification of their eligibility criteria by the research midwives at the academic hospital of Estaing or the clinical research assistants at the Vichy Hospital Center. If she is indeed eligible for the study, an inclusion visit will be scheduled. At this visit, the investigator-physician will verify the file with the woman (review her history) and examine the woman (blood pressure and examination of the skin of and around the scar). She will also receive a more detailed note of information. After a conversation with the investigator, who will answer her questions, the woman can sign the consent form. The investigator will also sign the consent form. The women will receive structured training on how to massage the scar (and also a paper information about the massage of the scar) and their first session of treatment by tecar therapy (or sham tecar therapy) at the end of this inclusion visit.

On average, the time to reflect between the first oral information about the study and the written consent signature will be one week.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman(≥18 years and ≤50 years), with a painful cesarean scar (VAS ≥ 4), at the 6-8 weeks postpartum visit (reimbursed by the French national health insurance fund), regardless of whether or not she is breastfeeding,
* Capable of providing informed consent to participate in this study,
* and affiliated with the French health insurance fund.

Exclusion Criteria:

* Refusal to participate,
* Has a pacemaker or a neurostimulator,
* Has an insulin pump,
* Coagulation disorders,
* Current thrombophlebitis,
* Current pregnancy,
* Burning sensation at the treatment area,
* Current cancer,
* Insensitivity to warm or to pain,
* Current infection (tuberculosis, etc.), especially of the surgical site,
* Current fever,
* Bladder wound during cesarean,
* Under guardianship or conservatorship, deprived freedom, or in the custody of correctional authorities,
* Keloid scar from previous cesarean,
* Previous tecar therapy,
* Strong hypertension (systolic > 150 or diastolic > 100) or hypotension (systolic ≤90 and diastolic < 40 mm Hg),
* Dermatologic lesion in the area to be treated (eczema, psoriasis, herpes zoster, etc.),
* subumbilical midline incision.
* Chronic inflammatory disease.
* Under a guardianship or conservatorship, deprived of freedom, or in the custody of correctional authorities.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Analgesic efficacy of tecar therapy on postoperative scar pain and/or discomfort | At 3 months after the cesarean delivery
  To study the analgesic efficacy of tecar therapy on postoperative scar pain and/or discomfort after cesarean delivery. Pain will be evaluated by a visual analogic scale (VAS) at 3 months post partum, by a ruler scored from 0 for no pain and/or discomfort to 10 for the worst imaginable.

SECONDARY OUTCOMES:
Pain and/or discomfort for cesarean scars at the end of all 3 sessions of tecar therapy | Week 3
  Pain and/or discomfort will be evaluated by a VAS, with a ruler scored from 0 for no pain to 10 for the worst imaginable.
Pain and/or discomfort due to cesarean scar at 6 months post partum | Month 6
  Pain and/or discomfort will be evaluated by a VAS, with a ruler scored from 0 for no pain to 10 for the worst imaginable.
Pain due to cesarean scar in the early postpartum period | Week 3
  Saint Antoine self-administered pain questionnaire, abridged version (QDSA, French adaptation of the McGill Pain questionnaire): at the end of the tecar therapy sessions
Pain due to cesarean scar in the early postpartum period | Month 3
  Saint Antoine self-administered pain questionnaire, abridged version (QDSA, French adaptation of the McGill Pain questionnaire): at the end of the tecar therapy sessions
Pain due to cesarean scar in the early postpartum period | Month 6
  Saint Antoine self-administered pain questionnaire, abridged version (QDSA, French adaptation of the McGill Pain questionnaire): at the end of the tecar therapy sessions
Pain due to cesarean scar in the early postpartum period | Week 3
  Self-administered brief pain questionnaire (QCD, French version of the "Brief Pain Inventory")
Pain due to cesarean scar in the early postpartum period | Month 3
  Self-administered brief pain questionnaire (QCD, French version of the "Brief Pain Inventory")
Pain due to cesarean scar in the early postpartum period | Month 6
  Self-administered brief pain questionnaire (QCD, French version of the "Brief Pain Inventory")
Research for neuropathic pain | Month 3
  Self-administered questionnaire to search for neuropathic pain [DN4]
Research for neuropathic pain | Month 6
  Self-administered questionnaire to search for neuropathic pain [DN4]
Interference with daily activities | Week 3
  Self-administered questionnaire "Multidimensional Pain Inventory" (MPI)
Interference with daily activities | Month 3
  Self-administered questionnaire "Multidimensional Pain Inventory" (MPI)
Interference with daily activities | Month 6
  Self-administered questionnaire "Multidimensional Pain Inventory" (MPI)
Anxiety and depression | Month 3
  Self-administered questionnaire "Hospital Anxiety and Depression Scale" (HADS)
Anxiety and depression | Month 6
  Self-administered questionnaire "Hospital Anxiety and Depression Scale" (HADS)
Health-related quality of life | Month 3
  self-administered questionnaire WHOQOL-BRIEF [WHO questionnaire on Quality of Life]
Health-related quality of life | Month 6
  self-administered questionnaire WHOQOL-BRIEF [WHO questionnaire on Quality of Life]
Quality of sexual life | Month 3
  Self-administered questionnaire "Female Sexual Function Index" [FSFI]
Quality of sexual life | Month 6
  Self-administered questionnaire "Female Sexual Function Index" [FSFI]
Quality of skin healing | Week 3
  Vancouver Scale
Consumption of analgesics or other co-treatments for analgesic purposes | During the 3 months of follow-up.
  consumption of analgesics and co-treatments collected prospectively during follow-up to allow the economic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Vendittelli, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No
The results generated by this research will be made available as soon as possible in an article. However, the individual data underlying the findings cannot be made freely available because of French legal restrictions. French Data Protection Agency (Commission Nationale de l'Informatique et des Libertés) accordingly strictly forbids making these data freely available. Nonetheless, aggregated anonymous data of the trial can be obtained upon request. Readers will be able to contact the corresponding author to request the data.

REFERENCES:
- [Derived] Grampayre M, Guiguet-Auclair C, Barasinski C, Vendittelli F. A sham-controlled randomised trial of Tecar therapy for painful caesarean scars: the NOCEPAIN study protocol. BMJ Open. 2025 Oct 6;15(10):e105743. doi: 10.1136/bmjopen-2025-105743. PMID 41057173